CLINICAL TRIAL: NCT01738048
Title: Persistent Pain After Reconstruction Following Mastectomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Danish Breast Cancer Cooperative Group (Other)
Responsible Party: Principal Investigator, Kenneth Geving Andersen, Physician, research fellow, Rigshospitalet, Denmark
Other Study IDs: H-D-2007-0099B
Record Dates: First submitted 2012-11-22; First posted 2012-11-30 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2012-11

CONDITIONS: Breast Cancer; Chronic Pain
Keywords: Pain; Neuropathic pain; Chronic pain
MeSH Terms: conditions — Breast Neoplasms; Chronic Pain; Pain; Neuralgia | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mastectomy: Patients treated with mastectomy without reconstruction
- Reconstruction: Patients treated with mastectomy followed by reconstruction
  Interventions: Procedure: Reconstruction

INTERVENTIONS:
Procedure: Reconstruction — Reconstructive surgery after mastectomy, either by expander or autologous tissue. Includes both primary and secondary reconstruction
  Groups: Reconstruction

SUMMARY:
A cross sectional study to determine the prevalence of persistent pain after reconstructive surgery after mastectomy for breast cancer, with a comparative analysis of a cohort treated with mastectomy without reconstruction.

DETAILED DESCRIPTION:
The aim of the study is to determine if reconstruction of the breast after mastectomy increases the risk of reporting persistent pain 2-3 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral primary breast cancer aged 18-70 years

Exclusion Criteria:

* recurrent cancer
* other malignancy
* emigration
* non-standardized treatment

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nationwide cross-sectional cohort
Sampling Method: Probability Sample
Enrollment: 1352 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
The risk of developing persistent if reconstructed | Cross-sectional, 2-3 years after surgery for breast cancer
  The risk of developing persistent if reconstructed compared to patients mastectomized without reconstruction expressed as an odds ratio.

SECONDARY OUTCOMES:
Prevalence of persistent pain after reconstruction after mastectomy | Cross-sectional, 2-3 years after surgery for breast cancer
  Self reported pain expressed as a percentage of the population of patients reconstructed with expander and autologous tissue. Pain intensity measured with a numerical rating scale 0-10, divided in mild (NRS 1-3), moderate (4-6) and severe pain (7-10). Patients regarded as having clinically relevant pain: NRS 4 or above, at least at a weekly basis.
Prevalence of sensory disturbances after reconstruction after mastectomy | Cross-sectional, 2-3 years after surgery for breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G Andersen, MD, Principal Investigator — Rigshospitalet, University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953